CLINICAL TRIAL: NCT04647383
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, 2-Period, Crossover Study to Evaluate the Respiratory Safety of Lemborexant in Adult and Elderly Subjects With Moderate to Severe Obstructive Sleep Apnea and Adult and Elderly Subjects With Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Evaluate the Respiratory Safety of Lemborexant in Adult and Elderly Participants With Moderate to Severe Obstructive Sleep Apnea, and in Adult and Elderly Participants With Moderate to Severe Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: E2006-A001-113
Record Dates: First submitted 2020-11-26; First posted 2020-11-30 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2022-02

CONDITIONS: Sleep Apnea, Obstructive; Pulmonary Disease, Chronic Obstructive; Respiration Disorders
Keywords: E2006; Lemborexant; Peripheral Oxygen Saturation; Apnea Hypopnea Index
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pulmonary Disease, Chronic Obstructive; Respiration Disorders | interventions — lemborexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- OSA Cohort, Sequence A: Placebo + Lemborexant 10 mg (Experimental): Participants with OSA will receive one lemborexant-matched placebo tablet on the night of Day 1 through Day 8 of Treatment Period 1, followed by one lemborexant 10 mg tablet on the night of Day 1 through Day 8 of Treatment Period 2. A washout period of 14 days will be maintained between the 2 treatment periods.
  Interventions: Drug: Placebo; Drug: Lemborexant 10 mg
- OSA Cohort, Sequence B: Lemborexant 10 mg + Placebo (Experimental): Participants with OSA will receive one lemborexant 10 mg tablet on the night of Day 1 through Day 8 of Treatment Period 1, followed by one lemborexant-matched placebo tablet on the night of Day 1 through Day 8 of Treatment Period 2. A washout period of 14 days will be maintained between the 2 treatment periods.
  Interventions: Drug: Placebo; Drug: Lemborexant 10 mg
- COPD Cohort, Sequence C: Placebo + Lemborexant 10 mg (Experimental): Participants with COPD will receive one lemborexant-matched placebo tablet on the night of Day 1 through Day 8 of Treatment Period 1, followed by one lemborexant 10 mg tablet on the night of Day 1 through Day 8 of Treatment Period 2. A washout period of 14 days will be maintained between the 2 treatment periods.
  Interventions: Drug: Placebo; Drug: Lemborexant 10 mg
- COPD Cohort, Sequence D: Lemborexant 10 mg + Placebo (Experimental): Participants with COPD will receive one lemborexant 10 mg tablet on the night of Day 1 through Day 8 of Treatment Period 1, followed by one lemborexant-matched placebo tablet on the night of Day 1 through Day 8 of Treatment Period 2. A washout period of 14 days will be maintained between the 2 treatment periods.
  Interventions: Drug: Placebo; Drug: Lemborexant 10 mg

INTERVENTIONS:
Drug: Placebo — OSA: Lemborexant-matched oral placebo will be administered at bedtime in the clinic (within 5 minutes before lights off) or at home when not in the clinic.
  Other Names: E2006
  Arms: OSA Cohort, Sequence A: Placebo + Lemborexant 10 mg; OSA Cohort, Sequence B: Lemborexant 10 mg + Placebo
Drug: Lemborexant 10 mg — OSA: 10 mg oral lemborexant will be administered at bedtime in the clinic (within 5 minutes before lights off) or at home when not in the clinic.
  Other Names: E2006
  Arms: OSA Cohort, Sequence A: Placebo + Lemborexant 10 mg; OSA Cohort, Sequence B: Lemborexant 10 mg + Placebo
Drug: Placebo — COPD: Lemborexant-matched oral placebo will be administered at bedtime in the clinic (within 5 minutes before lights off) or at home when not in the clinic.
  Other Names: E2006
  Arms: COPD Cohort, Sequence C: Placebo + Lemborexant 10 mg; COPD Cohort, Sequence D: Lemborexant 10 mg + Placebo
Drug: Lemborexant 10 mg — COPD: 10 mg oral lemborexant will be administered at bedtime in the clinic (within 5 minutes before lights off) or at home when not in the clinic.
  Other Names: E2006
  Arms: COPD Cohort, Sequence C: Placebo + Lemborexant 10 mg; COPD Cohort, Sequence D: Lemborexant 10 mg + Placebo

SUMMARY:
The primary purpose of the study is to determine whether lemborexant increases the apnea hypopnea index (AHI) on Day 8 of treatment in adult and elderly participants (adults greater than or equal to [>=] 45 to less than [<] 65 years; elderly >=65 to 90 years) with moderate to severe obstructive sleep apnea (OSA) compared with placebo, and using pulse oximetry determine whether lemborexant decreases the peripheral oxygen saturation (SpO2) during total sleep time (TST) on Day 8 of treatment in adult and elderly participants (adults >=45 to <65 years; elderly >=65 to 90 years) with moderate to severe chronic obstructive pulmonary disease (COPD) compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age >=45 and <=90 at the time of informed consent
2. Voluntary agreement and ability to provide written informed consent
3. Body mass index (BMI) <40 Kilogram per meter square (kg/m^2)
4. Reports habitually sleeping for at least 5.5 hours per night
5. Reports habitual bedtime between 21:00 and midnight
6. Agrees to stay in bed for 7 hours per night for the duration of the study
7. At Screening Visit 2: Has completed the sleep diary for at least 5 consecutive nights
8. At Screening Visit 2: Confirmation of mean habitual bedtime (MHB) between 21:00 and midnight (sleep diary)

   Additional Inclusion Criteria (OSA Cohort)
9. Moderate to severe OSA diagnosed according to the criteria of the ICSD, confirmed by PSG (home sleep testing by portable monitor is acceptable) within the previous 5 years or a repeated PSG during screening
10. On screening PSG: moderate OSA (defined as 15 <=AHI <30) or severe OSA (defined as AHI >=30 per hour)
11. SpO2 >=94% assessed as part of vital signs at Screening Visit 1

    Additional Inclusion Criteria (COPD Cohort)
12. Screening spirometry performed as per the Global Initiative for Obstructive Lung Disease (GOLD) recommendations
13. On screening spirometry, based on post-bronchodilator Forced Expiratory Volume in 1 second (FEV1):

    • FEV1/Forced Vital Capacity (FVC) <0.70 and one of the following:
    * 50% <=FEV1 <80% predicted (GOLD 2 Classification for moderate COPD) or
    * 30% <=FEV1 <50% predicted (GOLD 3 Classification for severe COPD)
14. Moderate to severe COPD according to medical history and screening spirometry as per the GOLD criteria (GOLD 2019)
15. On screening PSG

    * AHI <15
    * SpO2 during wakefulness >90% (both supine and sitting)
    * SpO2 during sleep >=80% for at least 75% of the recording period with no more than five continuous minutes <80% and with no SpO2 readings <70%

Exclusion Criteria:

1. Females of childbearing potential
2. A current diagnosis of restless legs syndrome, periodic limb movement disorder, circadian rhythm sleep disorder, or narcolepsy
3. Reports symptoms potentially related to narcolepsy, that in the clinical opinion of the investigator indicate the need for referral for a diagnostic evaluation for the presence of narcolepsy
4. A history of symptoms of rapid eye movement (REM) Behavior Disorder, sleep-related violent behavior, sleep-driving, or sleep-eating, or symptoms of another parasomnia that in the investigator's opinion make the participant unsuitable for the study
5. Periodic Limb Movement with Arousal Index (PLMAI) as measured on the screening

   PSG:
   * Age 18 to <65 years: PLMAI >=10
   * Age >65 years: PLMAI >15
6. A prolonged QT interval by Fredericia (QTcF) (QTcF >450 milliseconds [ms]) as demonstrated by a repeated electrocardiogram (ECG) at Screening
7. Any suicidal ideation with intent with or without a plan at Screening or within 6 months of Screening (that is, answering "Yes" to questions 4 or 5 on the Suicidal Ideation section of the Columbia-Suicide Severity Rating Scale [C-SSRS])
8. Any lifetime suicidal behavior (per the Suicidal Behavior section of the C-SSRS) within 10 years of Screening
9. Evidence of clinically significant disease (example, cardiac, respiratory, gastrointestinal, renal disease) that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments
10. Hypersensitivity to the study drug or any of the excipients
11. Used any prohibited prescription or over-the-counter medications within 1 week or 5 half-lives, whichever is longer, before the screening PSG
12. Any history of or concomitant medical condition that in the opinion of the investigator(s) would compromise the participant's ability to safely complete the study
13. Scheduled for surgery during the study that requires general anesthesia or administration of prohibited medications
14. Psychotic disorder(s) or unstable recurrent affective disorder(s) evident by use of antipsychotics or prior suicide attempt(s) within approximately the last 2 years
15. History of drug or alcohol dependency or abuse within approximately the last 2 years
16. Use of illegal recreational drugs (includes marijuana, regardless of whether prescribed for medicinal use)
17. Currently enrolled in another clinical study or used any investigational drug or device within 28 days or 5*the half-life, whichever is longer preceding informed consent
18. Previously participated in other clinical trial of lemborexant
19. Exposure within the last 14 days to an individual with confirmed or probable corona virus disease 2019 (COVID-19) or symptoms within the last 14 days that are on the most recent Centers for Disease Control and Prevention (CDC) list of COVID symptoms or any other reason to consider the participant at potential risk for an acute COVID-19 infection

    Additional Exclusion Criteria (OSA Cohort)
20. SpO2 <80% for >=5% of TST during the screening PSG
21. Use of a continuous positive airway pressure (CPAP) device or dental appliance within 2 weeks of the screening PSG, and does not agree to abstain from the use of a CPAP device or dental appliance from the
22. Current evidence of a clinically significant, active respiratory disorder other than OSA. This includes bronchiectasis, emphysema, asthma, COPD or any other pulmonary disorder identified by review of medical history, physical examination, and which in the opinion of the investigator, could compromise the participant's safety or interfere with study assessments
23. Current evidence of other clinically significant disease (example, psychiatric disorders, disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, cardiovascular system, or a congenital abnormality), malignancy within the past 5 years (other than adequately treated basal cell carcinoma or in situ carcinoma of the cervix), or chronic pain that in the opinion of the investigator could affect the participant's safety or interfere with the study assessments. Screening Visit through the last study visit

    Additional Exclusion Criteria (COPD Cohort)
24. Use of continuous (>16 hours/day) oxygen therapy
25. Use of oxygen therapy during PSG
26. Determination that, in the opinion of the investigator, removal of oxygen therapy could affect the participant's safety or interfere with the study assessments
27. Recent changes to COPD medications or recent acute exacerbation of COPD (that is, needing hospitalization or treatment with oral corticosteroids and/or antibiotics) within 3 months of enrollment
28. On screening spirometry (COPD only):

    * FEV1/FVC >=0.70
    * FEV1 >=80% predicted (GOLD 1 Classification for mild COPD)
    * FEV1 <30% predicted (GOLD 4 Classification for very severe COPD)
29. On screening PSG (COPD only):

    * Moderate to severe OSA (AHI >=15)
    * SpO2 <90% during wakefulness (supine and sitting)
    * SpO2 during sleep <80% for 25% or more of the recording with >5 consecutive minutes <80% and any SpO2 reading <70%
30. ECG evidence of right ventricular hypertrophy or right heart failure
31. Screening hematocrit >55%
32. Use of a CPAP device or dental appliance within 2 weeks of the screening PSG, and does not agree to abstain from the use of a CPAP device or dental appliance from the Screening Visit through the last study visit
33. Current evidence of a clinically significant, active respiratory disorder other than COPD and mild OSA. This includes any other pulmonary disorder identified by review of medical history, physical examination, and which in the opinion of the investigator, could compromise the participant's safety or interfere with study assessments.
34. Current evidence of other clinically significant disease other than COPD and mild OSA (example, psychiatric disorders, disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, cardiovascular system, or a congenital abnormality), malignancy within the past 5 years (other than adequately treated basal cell carcinoma or in situ carcinoma of the cervix), or chronic pain that in the opinion of the investigator could affect the participant's safety or interfere with the study assessments.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Pulmonary Associates, Glendale, Arizona
  - Pacific Research Network, San Diego, California
  - Teradan Clinical Trials, Brandon, Florida
  - St. Francis Medical Institute, Clearwater, Florida
  - Research Centers of America, Hollywood, Florida
  - Clinical Trials of Florida, LLC, Miami, Florida
  - Clinical Site Partners Orlando, LLC, Winter Park, Florida
  - NeuroTrials Research Inc., Atlanta, Georgia
  - GNP Research, Valdosta, Georgia
  - CTI Clinical Trial & Consulting Services, Cincinnati, Ohio
  - Intrepid Research, LLC, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

REFERENCES:
- [Derived] Khullar A, Boulos MI, Mak MSB, Moline M, Cheng JY, Hall N. Effect of lemborexant on sleep parameters and architecture in adult and elderly participants with mild-to-severe obstructive sleep apnea. Sleep Med. 2025 Oct;134:106757. doi: 10.1016/j.sleep.2025.106757. Epub 2025 Aug 18. PMID 40848323
- [Derived] Cheng JY, Lorch D, Hall N, Moline M. Respiratory safety of lemborexant in adult and elderly subjects with moderate-to-severe chronic obstructive pulmonary disease. J Sleep Res. 2025 Apr;34(2):e14334. doi: 10.1111/jsr.14334. Epub 2024 Sep 12. PMID 39266012
- [Derived] Cheng JY, Lorch D, Lowe AD, Uchimura N, Hall N, Shah D, Moline M. A randomized, double-blind, placebo-controlled, crossover study of respiratory safety of lemborexant in moderate to severe obstructive sleep apnea. J Clin Sleep Med. 2024 Jan 1;20(1):57-65. doi: 10.5664/jcsm.10788. PMID 37677076

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 10 investigative sites in the United States from 06 January 2021 to 10 February 2022.
Pre-assignment Details: A total of 48 participants for the obstructive sleep apnea (OSA) cohort were screened, of which 15 were screen failures and 33 were randomized in OSA cohort to receive study treatment. A total of 108 participants were screened for the chronic obstructive pulmonary disease (COPD) cohort, of which 78 were screen failures and 30 were randomized in COPD cohort to receive study treatment.
Groups:
- OSA Cohort, Sequence A: Placebo + Lemborexant 10 mg: Participants with OSA received lemborexant-matched placebo tablet, orally, once daily on the night (within 5 minutes of lights off) of Day 1 through Day 8 of Treatment Period 1, followed by lemborexant 10 milligram (mg) tablet, orally, once daily on the night (within 5 minutes of lights off) of Day 1 through Day 8 of Treatment Period 2. A washout period of 14 days was maintained between both treatment periods.
- OSA Cohort, Sequence B: Lemborexant 10 mg + Placebo: Participants with OSA received lemborexant 10 mg tablet, orally, once daily on the night (within 5 minutes of lights off) of Day 1 through Day 8 of Treatment Period 1, followed by one lemborexant-matched placebo tablet, orally, once daily on the night (within 5 minutes of lights off) of Day 1 through Day 8 of Treatment Period 2. A washout period of 14 days was maintained between both treatment periods.
- COPD Cohort, Sequence C: Placebo + Lemborexant 10 mg: Participants with COPD received lemborexant-matched placebo tablet, orally, once daily on the night (within 5 minutes of lights off) of Day 1 through Day 8 of Treatment Period 1, followed by lemborexant 10 mg tablet, orally, once daily on the night (within 5 minutes of lights off) of Day 1 through Day 8 of Treatment Period 2. A washout period of 14 days was maintained between both treatment periods.
- COPD Cohort, Sequence D: Lemborexant 10 mg + Placebo: Participants with COPD received lemborexant 10 mg tablet, orally, once daily on the night (within 5 minutes of lights off) of Day 1 through Day 8 of Treatment Period 1, followed by lemborexant-matched placebo tablet, orally, once daily on the night (within 5 minutes of lights off) of Day 1 through Day 8 of Treatment Period 2. A washout period of 14 days was maintained between both treatment periods.
Period: Treatment Period 1 (8 Days)
Arm/Group | OSA Cohort, Sequence A: Placebo + Lemborexant 10 mg | OSA Cohort, Sequence B: Lemborexant 10 mg + Placebo | COPD Cohort, Sequence C: Placebo + Lemborexant 10 mg | COPD Cohort, Sequence D: Lemborexant 10 mg + Placebo
Started | 16 | 17 | 14 | 16
Completed | 16 | 17 | 14 | 16
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period (14 Days)
Arm/Group | OSA Cohort, Sequence A: Placebo + Lemborexant 10 mg | OSA Cohort, Sequence B: Lemborexant 10 mg + Placebo | COPD Cohort, Sequence C: Placebo + Lemborexant 10 mg | COPD Cohort, Sequence D: Lemborexant 10 mg + Placebo
Started | 16 | 17 | 14 | 16
Completed | 16 | 17 | 14 | 16
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2 (8 Days)
Arm/Group | OSA Cohort, Sequence A: Placebo + Lemborexant 10 mg | OSA Cohort, Sequence B: Lemborexant 10 mg + Placebo | COPD Cohort, Sequence C: Placebo + Lemborexant 10 mg | COPD Cohort, Sequence D: Lemborexant 10 mg + Placebo
Started | 16 | 17 | 14 | 16
Completed | 16 | 16 | 14 | 16
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set for each cohort was the group of participants who received at least 1 dose of study drug and had at least 1 post-dose safety assessment.
Groups:
- OSA Cohort, Sequence A: Placebo + Lemborexant 10 mg: Participants with OSA received lemborexant-matched placebo tablet, orally, once daily on the night (within 5 minutes of lights off) of Day 1 through Day 8 of Treatment Period 1, followed by lemborexant 10 mg tablet, orally, once daily on the night (within 5 minutes of lights off) of Day 1 through Day 8 of Treatment Period 2. A washout period of 14 days was maintained between both treatment periods.
- Total: Total of all reporting groups
Arm/Group | OSA Cohort, Sequence A: Placebo + Lemborexant 10 mg | OSA Cohort, Sequence B: Lemborexant 10 mg + Placebo | COPD Cohort, Sequence C: Placebo + Lemborexant 10 mg | COPD Cohort, Sequence D: Lemborexant 10 mg + Placebo | Total
Number analyzed (Participants) | 16 | 17 | 14 | 16 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 3 | 4 | 29
  >=65 years | 5 | 6 | 11 | 12 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 11 | 10 | 31
  Male | 13 | 10 | 3 | 6 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 2 | 2 | 11
  Not Hispanic or Latino | 11 | 15 | 12 | 14 | 52
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 12 | 13 | 14 | 51
  Black or African American | 3 | 4 | 1 | 2 | 10
  Japanese | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: OSA Cohort: Apnea-Hypopnea Index (AHI) on Day 8 of Treatment Periods 1 and 2
Description: AHI was the number of apneas and hypopneas divided by the total sleep time (TST) (in minutes) and multiplied by 60 (minute per hour [min/hour]) (that is, the average number of apneas and hypopneas per hour of sleep), as defined by the American Academy of Sleep Medicine. An AHI greater than or equal to (>=) 5 to less than (<) 15 is classed as mild, AHI >=15 to <30 as moderate, and AHI >=30 as severe. TST was defined as the total time asleep in minutes using polysomnography (PSG).
Time Frame: Day 8 of Treatment Periods 1 and 2 (up to Day 30)
Population: The pharmacodynamic (PD) analysis set for each cohort was the group of participants who had sufficient PD data to derive at least 1 primary PD parameter. Here, "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: events (apnea plus hyponea) per hour
Groups:
- OSA Cohort: Placebo: Participants with OSA received lemborexant-matched placebo tablet, orally, once daily on the night (within 5 minutes of lights off) of Day 1 through Day 8 of Treatment Periods 1 and 2. A washout period of 14 days was maintained between both treatment periods.
- OSA Cohort: Lemborexant 10 mg: Participants with OSA received lemborexant 10 mg tablet, orally, once daily on the night (within 5 minutes of lights off) of Day 1 through Day 8 of Treatment Periods 1 and 2. A washout period of 14 days was maintained between both treatment periods.
Arm/Group | OSA Cohort: Placebo | OSA Cohort: Lemborexant 10 mg
Number analyzed (Participants) | 32 | 33
events (apnea plus hyponea) per hour | 45.09 (22.851) | 44.90 (22.246)

2. Primary Outcome: COPD Cohort: Peripheral Oxygen Saturation (SpO2) During TST on Day 8 of Treatment Periods 1 and 2
Description: SpO2 is an estimate of the amount of oxygen in the blood. It is the percentage of hemoglobin containing oxygen compared to the total amount of hemoglobin in the blood (that is, oxygenated hemoglobin versus oxygenated and non-oxygenated hemoglobin). SpO2 was monitored by noninvasive method known as transmissive pulse oximetry. TST was defined as the total time asleep in minutes using PSG.
Time Frame: Day 8 of Treatment Periods 1 and 2 (up to Day 30)
Population: The PD analysis set for each cohort was the group of participants who had sufficient PD data to derive at least 1 primary PD parameter.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Groups:
- COPD Cohort: Placebo: Participants with COPD received lemborexant-matched placebo tablet, orally, once daily on the night (within 5 minutes of lights off) of Day 1 through Day 8 of Treatment Periods 1 and 2. A washout period of 14 days was maintained between both treatment periods.
- COPD Cohort: Lemborexant 10 mg: Participants with COPD received lemborexant 10 mg tablet, orally, once daily on the night (within 5 minutes of lights off) of Day 1 through Day 8 of Treatment Periods 1 and 2. A washout period of 14 days was maintained between both treatment periods.
Arm/Group | COPD Cohort: Placebo | COPD Cohort: Lemborexant 10 mg
Number analyzed (Participants) | 30 | 30
percentage of oxygen saturation | 90.80 (2.565) | 91.27 (2.227)

3. Secondary Outcome: OSA Cohort: AHI on Day 1 of Treatment Periods 1 and 2
Description: AHI was the number of apneas and hypopneas divided by the TST (in minutes) and multiplied by 60 (min/hour) (that is, the average number of apneas and hypopneas per hour of sleep), as defined by the American Academy of Sleep Medicine. An AHI >=5 to <15 is classed as mild, >=15 to <30 as moderate, and AHI >=30 as severe. TST was defined as the total time asleep in minutes using PSG.
Time Frame: Day 1 of Treatment Periods 1 and 2 (up to Day 23)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: events (apnea plus hyponea) per hour
Arm/Group | OSA Cohort: Placebo | OSA Cohort: Lemborexant 10 mg
Number analyzed (Participants) | 33 | 33
events (apnea plus hyponea) per hour | 44.65 (25.770) | 41.64 (21.215)

4. Secondary Outcome: OSA Cohort: Peripheral SpO2 During TST on Days 1 and 8 of Treatment Periods 1 and 2
Description: as for outcome 2
Time Frame: Days 1 and 8 of Treatment Periods 1 and 2 (up to Day 30)
Population: The PD analysis set for each cohort was the group of participants who had sufficient PD data to derive at least 1 primary PD parameter. Here, "number analyzed" signifies those participants who were evaluable at given timepoint for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | OSA Cohort: Placebo | OSA Cohort: Lemborexant 10 mg
Number analyzed (Participants) | 33 | 33
percentage of oxygen saturation
  Day 1 | 93.12 (2.073) | 93.00 (2.462)
  Day 8: number analyzed (Participants) | 32 | 33
  Day 8 | 93.44 (1.983) | 93.06 (1.983)

5. Secondary Outcome: OSA Cohort: Percentage (%) of TST During Which SpO2 Was <90%, <85% and <80% on Days 1 and 8 of Treatment Periods 1 and 2
Description: TST was defined as the total time asleep in minutes using PSG. SpO2 is an estimate of the amount of oxygen in the blood. It is the percentage of hemoglobin containing oxygen compared to the total amount of hemoglobin in the blood (that is, oxygenated hemoglobin versus oxygenated and non-oxygenated hemoglobin). SpO2 was monitored by noninvasive method known as transmissive pulse oximetry.
Time Frame: Days 1 and 8 of Treatment Periods 1 and 2 (up to Day 30)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of TST
Arm/Group | OSA Cohort: Placebo | OSA Cohort: Lemborexant 10 mg
Number analyzed (Participants) | 33 | 33
percentage of TST
  Day 1: SpO2 <90% | 11.966 (16.8941) | 12.849 (15.5993)
  Day 1: SpO2 <85% | 2.708 (4.9400) | 3.748 (6.6010)
  Day 1: SpO2 <80% | 0.776 (1.7896) | 1.125 (2.5021)
  Day 8: SpO2 <90%: number analyzed (Participants) | 32 | 33
  Day 8: SpO2 <90% | 9.474 (9.7930) | 11.295 (12.6345)
  Day 8: SpO2 <85%: number analyzed (Participants) | 32 | 33
  Day 8: SpO2 <85% | 2.283 (3.6302) | 2.696 (4.4283)
  Day 8: SpO2 <80%: number analyzed (Participants) | 32 | 33
  Day 8: SpO2 <80% | 0.522 (1.3345) | 0.651 (1.3153)

6. Secondary Outcome: OSA Cohort: Mean Oxygen Desaturation Index (ODI) on Days 1 and 8 of Treatment Periods 1 and 2
Description: ODI was defined as (oxygen desaturations >=3%*60)/TST (that is, the average number of oxygen desaturations >=3% per hour of sleep), as defined by the American Academy of Sleep Medicine. TST was defined as the total time asleep in minutes using PSG.
Time Frame: Days 1 and 8 of Treatment Periods 1 and 2 (up to Day 30)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | OSA Cohort: Placebo | OSA Cohort: Lemborexant 10 mg
Number analyzed (Participants) | 33 | 33
events per hour
  Day 1 | 39.71 (24.547) | 36.52 (20.325)
  Day 8: number analyzed (Participants) | 32 | 33
  Day 8 | 39.07 (21.475) | 39.51 (22.037)

7. Secondary Outcome: OSA Cohort: Absolute Number of Desaturations (>=3% Reduction From Baseline SpO2) on Days 1 and 8 of Treatment Periods 1 and 2
Description: Desaturation was defined as decrease in the mean SpO2 of >=3% (over the last 120 seconds) that lasts for at least 10 seconds. SpO2 is an estimate of the amount of oxygen in the blood. It is the percentage of hemoglobin containing oxygen compared to the total amount of hemoglobin in the blood (that is, oxygenated hemoglobin versus oxygenated and non-oxygenated hemoglobin). SpO2 was monitored by noninvasive method known as transmissive pulse oximetry.
Time Frame: Days 1 and 8 of Treatment Periods 1 and 2 (up to Day 30)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: events (number of desaturations)
Arm/Group | OSA Cohort: Placebo | OSA Cohort: Lemborexant 10 mg
Number analyzed (Participants) | 33 | 33
events (number of desaturations)
  Day 1 | 253.85 (161.971) | 256.52 (141.952)
  Day 8: number analyzed (Participants) | 32 | 33
  Day 8 | 255.28 (149.158) | 273.97 (155.209)

8. Secondary Outcome: COPD Cohort: Peripheral SpO2 During TST on Day 1 of Treatment Periods 1 and 2
Description: as for outcome 2
Time Frame: Day 1 of Treatment Periods 1 and 2 (up to Day 23)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | COPD Cohort: Placebo | COPD Cohort: Lemborexant 10 mg
Number analyzed (Participants) | 30 | 30
percentage of oxygen saturation | 91.53 (2.161) | 91.13 (2.801)

9. Secondary Outcome: COPD Cohort: AHI on Days 1 and 8 of Treatment Periods 1 and 2
Description: as for outcome 3
Time Frame: Days 1 and 8 of Treatment Periods 1 and 2 (up to Day 30)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: events (apnea plus hyponea) per hour
Arm/Group | COPD Cohort: Placebo | COPD Cohort: Lemborexant 10 mg
Number analyzed (Participants) | 30 | 30
events (apnea plus hyponea) per hour
  Day 1 | 6.09 (4.827) | 7.40 (6.331)
  Day 8 | 5.88 (5.245) | 6.15 (5.185)

10. Secondary Outcome: COPD Cohort: Percentage of TST During Which SpO2 Was <90%, <85% and <80% on Days 1 and 8 of Treatment Periods 1 and 2
Description: as for outcome 5
Time Frame: Days 1 and 8 of Treatment Periods 1 and 2 (up to Day 30)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of TST
Arm/Group | COPD Cohort: Placebo | COPD Cohort: Lemborexant 10 mg
Number analyzed (Participants) | 30 | 30
percentage of TST
  Day 1: SpO2 <90% | 15.593 (23.3552) | 21.468 (30.0042)
  Day 1: SpO2 <85% | 0.860 (1.9286) | 3.286 (9.0190)
  Day 1: SpO2 <80% | 0.155 (0.5416) | 0.224 (0.5912)
  Day 8: SpO2 <90% | 22.991 (30.9595) | 21.086 (30.3560)
  Day 8: SpO2 <85% | 3.330 (9.9935) | 1.151 (3.1124)
  Day 8: SpO2 <80% | 0.152 (0.4743) | 0.075 (0.2218)

11. Secondary Outcome: COPD Cohort: Mean ODI on Days 1 and 8 of Treatment Periods 1 and 2
Description: as for outcome 6
Time Frame: Days 1 and 8 of Treatment Periods 1 and 2 (up to Day 30)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | COPD Cohort: Placebo | COPD Cohort: Lemborexant 10 mg
Number analyzed (Participants) | 30 | 30
events per hour
  Day 1 | 4.61 (4.462) | 5.46 (4.823)
  Day 8 | 4.34 (4.562) | 4.71 (4.772)

12. Secondary Outcome: COPD Cohort: Absolute Number of Desaturations (>=3% Reduction From Baseline SpO2) on Days 1 and 8 of Treatment Periods 1 and 2
Description: as for outcome 7
Time Frame: Days 1 and 8 of Treatment Periods 1 and 2 (up to Day 30)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: events (number of desaturations)
Arm/Group | COPD Cohort: Placebo | COPD Cohort: Lemborexant 10 mg
Number analyzed (Participants) | 30 | 30
events (number of desaturations)
  Day 1 | 26.77 (27.485) | 36.07 (31.509)
  Day 8 | 25.33 (28.243) | 29.97 (33.055)

ADVERSE EVENTS:
Time Frame: Baseline up to end of follow up visit (up to 59 days)
Arm/Group | OSA Cohort: Placebo | OSA Cohort: Lemborexant 10 mg | COPD Cohort: Placebo | COPD Cohort: Lemborexant 10 mg
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/33 | 0/33 | 0/30 | 1/30
Other Adverse Events (participants affected / at risk) | 0/33 | 2/33 | 2/30 | 1/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OSA Cohort: Placebo (N=33) | OSA Cohort: Lemborexant 10 mg (N=33) | COPD Cohort: Placebo (N=30) | COPD Cohort: Lemborexant 10 mg (N=30)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OSA Cohort: Placebo (N=33) | OSA Cohort: Lemborexant 10 mg (N=33) | COPD Cohort: Placebo (N=30) | COPD Cohort: Lemborexant 10 mg (N=30)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT04647383/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/83/NCT04647383/SAP_001.pdf